CLINICAL TRIAL: NCT05062967
Title: Evaluation of Orthohepevirus C Infection as an Emerging Cause of Zoonotic Origin Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: PI21/00793
Record Dates: First submitted 2021-09-17; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis; Liver Diseases; Acute Hepatitis; Chronic Hepatitis; Liver Disease Chronic
Keywords: Orthohepevirus C; Hepatitis; Liver Diseases
MeSH Terms: conditions — Hepatitis; Liver Diseases; Hepatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- HAOD Cohort: This cohort includes patients with acute hepatitis of unknown origin, meaning its origin could not be determined after screening of (at least) HAV, HAB, HAC, HAE, Epstein-Barr virus and cytomegalovirus. Patients will be recruited in 17 centres nationwide.
  The research group will receive a 1mL plasma / serum sample from each patient to study the presence of Ortho-C infection
- OrthoC-Tx Cohort: This cohort includes liver or kidney transplant patients under follow-up. The research group will receive a 1mL plasma / serum sample every year from each patient to study the presence of Ortho-C infection
- Ortho-CoRIS Cohort: This cohort includes VIH positive patients who are in follow-up by the Spanish Network of AIDS Research.
  The research group will receive a plasma / serum sample every year from each patient to study the presence of Ortho-C infection.
- TrazHE Cohort: This cohort includes patients whose clinical picture is compatible with HAE infection.
  The presence of Ortho-C infection will be studied in patients with positive IgM for HAE and absence of RNA-HAE.
- Ortho-C-Rodent Cohort: This cohort includes wild rats. Feces and liver samples will be taken in order to determine the prevalence of Ortho-C in wild rats (Ortho-C's main reservoir).
- Ortho-C-Domestic Rodent Cohort: This cohort includes domestic rats and mustelids. Feces and liver samples will be taken in order to determine the prevalence of Ortho-C in domestic rats and mustelids.
- Ortho-C-Carnivore Cohort: This cohort includes 236 wild carnivores that feed off rodents. Carnivores' cause of death is they were run over.
  Feces, liver and serum samples will be taken to study the transmission of Ortho-C.

SUMMARY:
The main objective of this study is to evaluate the prevalence and the clinical impact of Orthohepevirus C infection in different human populations, and to determine its zoonotic origin comparing the sequences obtained in both human and animal populations. This is an ambispective study where Orthohepevirus C infection will be evaluated in four high risk human population: i) patients with acute hepatitis, ii) patients with positive IgM antibody against Hepatitis E virus infection with undetectable viral load, iii) HIV infected individuals, and iv) solid organ transplant recipients. Furthermore, we will analyze three animal populations: i) suburban rodents, ii) domestic rodents, iii) wild carnivores. Viral sequences identified in both human and animal populations will be compared to evaluate the zoonotic origin of the infections.

DETAILED DESCRIPTION:
To carry out the project a database will be created in electronic format, where the study team will integrate epidemiological, clinical and laboratory tests data of patients. Data will be anonymous and coded by a data manager.

Primary objective is to assess the prevalence of Ortho-C infection in patients with acute hepatitis of no identified origin

Secondary objectives are:

1. To evaluate the prevalence and risk factors of Ortho-C infection in patients with solid organ transplant.
2. To evaluate the prevalence and risk factors of Ortho-C infection in patients with HIV infection.
3. To assess the presence of Ortho-C infection in patients with the presence of antibodies (IgM) against HEV and absence of HEV-RNA
4. To evaluate the prevalence of infection by Ortho-C in wild and periurban rodents.
5. To evaluate the prevalence of infection by Ortho-C in domestic rodents and mustelids.
6. To evaluate the prevalence of infection by Ortho-C in wild carnivores
7. To molecularly characterize and evaluate the degree of homology of Ortho-C viral sequences found in humans and animals

ELIGIBILITY:
1. HAOD cohort (Cohort of patients with acute hepatitis of unknown origin)

* Patients older than 18 years with acute hepatitis of unknown origin (HAOD)

  2. OrthoC-Tx cohort (HEV Screening Cohort in Transplant Patients):
* Kidney or liver transplant subjects

  3. Ortho-CoRIS Cohort (derived from the AIDS Research Network Cohort (CoRIS))
* HIV-infected patients being monitored by the Spanish AIDS Research Network (RIS)

  4. TrazHE Cohort (Traceability cohort of Hepatitis E infections)
* Patients with the presence of antibodies (IgM) against HEV and absence of HEV-RNA

  5. Ortho-C-Rodent Collection:
* Wild and peri-urban rodents (rats) from different areas of Spain

  6. Ortho-C-Domestic Rodent Collection:
* Domestic rodents and mustelids under follow-up in veterinary clinics of different Spanish municipalities.

  7. Ortho-C-Carnivore Collection:
* Wild carnivores that eat rodents collected by the research team since 2020 in 4 autonomous communities (Extremadura, Andalusia, Murcia and Castilla la Mancha)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Depending on the cohort. Please see "Group and Interventions" section to learn about the study population in each cohort.
Sampling Method: Probability Sample
Enrollment: 3257 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Existence of Ortho-C infection | Yearly, up to three years.
  The presence of Ortho-C infection is defined by:
  * HAOD, TrazHE, OrthoC-Tx and Ortho-CoRIS cohorts: presence of RNA-OrthoC in blood.
  * Ortho-C-Rodent and Ortho-C-Carnivore cohorts: presence of RNA-OrthoC in serum, feces and/or liver tissue
  * Ortho-C-Domestic-Rodent cohort: presence of RNA-OrthoC in feces.

CONTACTS AND LOCATIONS:
Overall Officials: ANTONIO RIVERO ROMÁN, Principal Investigator — Hospital Universitario Reina Sofía
Locations (10):
- Spain (10):
  - Hospital de Jerez de La Frontera, Jerez de la Frontera, Cádiz
  - Hospital de Puerto Real, Puerto Real, Cádiz
  - Fundacion Instituto de Investigacion Sanitaria de Santiago de Compostela, Santiago de Compostela, Galicia
  - Instituto de Investigacion En Recursos Cinegeticos (Irec), Ciudad Real
  - Facultad de Veterinaria de Cordoba, Córdoba
  - Fundacion Investigacion Biomedica de Cordoba (Fibico), Córdoba
  - Instituto Maimonides de Investigacion Biomedica de Cordoba (Imibic), Córdoba
  - Hospital Universitario San Cecilio, Granada
  - Clinica Universidad de Navarra, Madrid
  - Complejo Hospitalario de Especialidades Virgen de La Victoria, Málaga

IPD SHARING:
Plan to Share IPD: Yes
Sharing the results of this study after they are made public.
Time Frame: After study results are published.
Access Criteria: Send access request to principal investigator.

REFERENCES:
- [Derived] Caballero-Gomez J, Casares-Jimenez M, Gallo-Marin M, Pereira-Pardo S, Beato-Benitez A, Poyato A, Guerra R, Avellon A, Schilling-Loeffler K, Freyre-Carrillo C, Garcia-Bocanegra I, Jimenez-Martin D, Corona-Mata D, Viciana I, Fajardo T, Munoz-Chimeno M, Quevedo MA, Rios-Munoz L, Perez AB, Cano-Terriza D, Macias J, Fuentes A, Johne R, Rivero-Juarez A, Rivero A; GEHEP-014 Study Group. Rat hepatitis E virus as an aetiological agent of acute hepatitis of unknown origin. J Hepatol. 2025 Sep;83(3):662-669. doi: 10.1016/j.jhep.2025.02.027. Epub 2025 Feb 26. PMID 40020930